CLINICAL TRIAL: NCT02831595
Title: Effectiveness of Titanium Niobium Nitride Coating in Total Knee Arthroplasty
Status: Terminated | Type: Observational
Why Stopped: Enrollment stopped for missing availability of the site
Sponsor: Permedica spa (Industry)
Responsible Party: Sponsor
Other Study IDs: VCG-30-2015
Record Dates: First submitted 2016-06-29; First posted 2016-07-13 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Knee Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients undergoing unilateral TKA
  Interventions: Device: GKS Prime Flex Bioloy by Permedica, a TiNbN coated fixed-bearing cruciate-retaining total knee prosthesis

INTERVENTIONS:
Device: GKS Prime Flex Bioloy by Permedica, a TiNbN coated fixed-bearing cruciate-retaining total knee prosthesis

SUMMARY:
Modern knee implants combine several types of metal and therefore potentially expose patients to different metal ions.

Titanium niobium nitride coating (TiNbN) acts like a physical barrier against the corrosion process and the metallic ions release towards the surrounding biologic environment, thus, making TiNbN-coated prostheses possible to be safety implanted in metal sensitized patients.

The aim of the study is to verify that the postoperative plasma metal concentrations at 1 year are not different than preoperative values.

ELIGIBILITY:
Inclusion Criteria:

* Patients candidate for unilateral primary total knee arthroplasty

Exclusion Criteria:

* Existing orthopaedic metal implants
* A history of hypersensitivity to metals
* Preoperative patch-test positivity to Co, Cr, Ni and Ti
* Malignancies
* Renal insufficiency
* Severe illnesses that would impair participation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of knee osteoarthritis scheduled for unilateral TKA
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-06; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline plasma metal ion concentrations (Co, Cr, Ni) at 12 months | Preoperative and at 12 months follow-up

SECONDARY OUTCOMES:
Number of patients with metal sensitivity at 1 year tested by patch-testing | 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Ursino, MD, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi Milano, Italy